CLINICAL TRIAL: NCT06474104
Title: Collection of Blood and Skin Samples From Patients With Primary Mitochondrial Diseases and Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MNV-008
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Primary Mitochondrial Diseases
Keywords: Mitochondrial; Research; PMD; Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Mitochondrial diseases are a genetically diverse group of disorders, some of which are caused by mutations or deletions in the mitochondrial DNA (mtDNA) and which display a wide range of severity and phenotypes. Despite a prevalence of roughly 1 in 8500 in the population there is no effective treatments for the majority of mitochondrial diseases beyond supportive care (Gorman 2016, Elliott 2008). Many of these, such as Pearson syndrome and Kearns-Sayre syndrome, are early onset disorders, and may lead to mortality within the first decades of life. Importantly, mitochondria are selectively inherited from the mother. In addition, there are numerous diseases in which mitochondrial dysfunction plays an important role. Some examples are Alzheimer's and Parkinson's disease, both of which are known to have mitochondrial involvement.

Minovia therapeutics develops a therapeutic intervention called mitochondrial augmentation technology (MAT). For the development work, Minovia needs patients' cells with different mutations that will allow to study the baseline heteroplasmy and functionality of patient hematopoietic cells, identify potential biomarkers to assess mitochondrial content and function in liquid biopsies, and study the efficacy of MAT in different PMDs.

DETAILED DESCRIPTION:
The aim of this study is to identify mitochondria-related potential biomarkers from peripheral blood specimens that will function as a diagnostic tool. The intention is to develop direct and indirect functional evaluation for mitochondria performance, and to perform a comparison analysis between healthy population and patients with compromised mitochondrial function. In order to define what is a dysfunctional mitochondrial with a clinical significance, the above assays will function as a junction between the mitochondria characteristics (i.e content and metabolic function) and the blood cell functionality, in order to both differentiate between the two cohorts by means of clinical correlation, as well as to set a clinical range that correlates to a pathology.

In addition, the study aims to gain a deeper understanding of the correlation between heteroplasmy level in different hematopoietic subsets in the different PMDs, and how this differential heteroplasmy may affect biomarker readouts and/or cell functionality or distribution.

In addition, this study aims to collect skin fibroblasts from PMD patients, for the purpose of establishing iPSC lines with different mtDNA mutations and/or deletions, in order to study efficacy of MAT in patient cells in pre-clinical models derived from these iPSC lines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 3 to 85 years.
2. For patients with Primary Mitochondrial Disease:

   a. Clinical diagnosis of PMD confirmed by mtDNA sequencing.
3. For Healthy Volunteers:

   1. Normal Vital signs and BMI for age
   2. No active medical conditions or diseases
   3. No current medications, other than acetaminophen and naproxen sodium
4. For All Subjects:

   1. No viral or bacterial illness in past 2 weeks
   2. No antibiotic or antiviral medications in past 2 weeks
   3. No blood transfusion in past 2 weeks
   4. No current pregnancy
   5. Not currently breastfeeding
   6. Alcohol use less than 2 drinks / day
   7. No recreational or illicit drug use in previous 1 year
   8. No tobacco or nicotine containing products in previous 1 year
5. Patient, parent or guardian able to understand and provide voluntary written informed consent.

Exclusion Criteria:

1. History of prior treatment with allogeneic hematopoietic stem cell transplantation, or gene therapy.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Samples of peripheral blood will be collected from up to 50 patients with PMD and up to 50 healthy volunteers.
  Samples of skin will be collected from up to 50 patients with PMD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
mitochondrial function | 1 year
  Analysis on how different mitochondrial mutations (sequence / heteroplasmy) are related to mitochondrial function and quantity in the white cell line and their characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center - Tel Ashomer, Ramat Gan, Israel, Israel